CLINICAL TRIAL: NCT02983994
Title: Errors in the Use of Turbuhaler and Spiromax Devices Patients With Asthma
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: FPS-INH-2016-01
Record Dates: First submitted 2016-11-23; First posted 2016-12-06 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2017-10

CONDITIONS: Asthma
Keywords: asthma, devices
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with asthma with an inhaled steroid: Patients with a diagnosis of asthma with indication of Treatment with an inhaled steroid (CI)
  Interventions: Device: TURBUHALER®
- Patients with asthma with an inhaled Beta agonist: Patients with a diagnosis of asthma with indication of Treatment with an inhaled Beta agonist (LABA)
  Interventions: Device: SPIROMAX®

INTERVENTIONS:
Device: TURBUHALER®
  Groups: Patients with asthma with an inhaled steroid
Device: SPIROMAX®
  Groups: Patients with asthma with an inhaled Beta agonist

SUMMARY:
The aim of the study is to evaluate the errors that may occur during inhalation of two devices in patients with asthma, as well as to study whether it relates to the degree of control of patient symptoms and the degree of compliance of medication symptoms. Finally, we also want to study the degree of patient satisfaction with each of the inhalers studied

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma with treatment indication with CI + LABA according to GINA 2015 guide and in dry powder device.
* Over 18 years.
* Patient in stable phase without having had exacerbations in the 3 months previous to the Inclusion in the study

Exclusion Criteria:

* Presence of relevant respiratory disease other than asthma (including COPD).
* Refusal to participate in the study and sign informed consent or inability to To give informed consent.
* Patients who have previously been treated with inhaled dust devices dry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as asthma with indication for treatment with an inhaled steroid (IC) and long-acting beta agonist (LABA), over 18 years of age, will be consecutively included according to the criteria of the GINA 2015 (Global Strategy for Asthma Management and Prevention), who have never used dry-powder inhalers, and whose doctor has prescribed one of the inhalation systems to be studied in the normal practice of the consultation. Patients will be recruited consecutively to complete the sample size established with each type of device, in each of the participating centers.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-11; Primary Completion 2017-05 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
The effectiveness of inhaler management. | two months
  The effectiveness of inhaler management, It will be the comparison of the means of the number of errors detected between both devices.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Regional de Málaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville